CLINICAL TRIAL: NCT04804514
Title: Phase 1/2a Study of KH001 in Dentin Hypersensitivity Patients
Brief Title: Evaluation of the Safety and Tolerability of KH001 in Dentin Hypersensitivity Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HysensBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KH001sol-01
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dentin Sensitivity
Keywords: Dentin regeneration; Hypersensitivity; Sensitivity; Tooth sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KH001 (Experimental): The study consists of sequential dosing cohorts, 8 subjects per cohort will be administered KH001 or placebo.
  Interventions: Drug: KH001
- Placebo (Placebo Comparator): The study consists of sequential dosing cohorts, 8 subjects per cohort will be administered KH001 or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KH001 — The study drug is applied to teeth
  Arms: KH001
Drug: Placebo — The placebo is applied to teeth
  Arms: Placebo

SUMMARY:
This is a phase 1/2a study in dentin hypersensitivity patients to assess the safety, tolerability, efficacy and pharmacokinetics of single and multiple doses of KH001.

ELIGIBILITY:
[Inclusion criteria]

1. Subjects must be fully aware of the purpose and the content of the study, and the characteristics of the Investigational Product to sign written consent of their free will to take part in the study;
2. Subjects having at least 20 natural teeth and two teeth that could be assessed
3. Subjects is diagnosed with dentin hypersensitivity, has experienced dental symptoms of two or more teeth

[Exclusion criteria]

1. Subjects is allergic to the active substance or other excipients used in the Investigational Product
2. Subjects has any history of clinically significant allergy, such as drug allergy, asthma, eczema, or anaphylaxis
3. Subjects has any disease related to dentin hypersensitivity
4. Subjects taking anti-inflammatory analgesic drugs

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events(AEs) | up to 22 days and 36 days
  The safety and tolerability of KH001 single and multiple ascending dose are evaluated.
  Adverse event(AE) is based on abnormal clinical laboratory tests, physical exam results and other medically assessments

SECONDARY OUTCOMES:
Change from baseline in VAS(Visual Analogue Score). | up to 22 days and 36 days
  VAS scale (0-100mm)
Maximum plasma concentration (Cmax) of KH001 single and multiple ascending dose. | 0~24 hours
  Pharmacokinetics parameter derived from plasma
Area under the concentration-time curve (AUC) of KH001 single and multiple ascending dose | 0~24 hours
  Pharmacokinetics parameter derived from plasma
Time to reach maximum concentration (Tmax) of KH001 single and multiple ascending dose | 0~24 hours
  Pharmacokinetics parameter derived from plasma
Elimination half life (t½) of KH001 single and multiple ascending dose | 0~24 hours
  Pharmacokinetics parameter derived from plasma
Estimate of apparent clearance (CL/F) of KH001 single and multiple ascending dose | 0~24 hours
  Pharmacokinetics parameter derived from plasma
Change from Baseline in Evaporative Air Sensitivity and Tactile Threshold | up to 22 days and 36 days
  pain intensity assessed by 0-3 scale
Change from baseline in Dentine Hypersensitivity Experience Questionnaire | up to 22 days and 36 days
  assessed by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Dental Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
HysensBio Inc. will not be sharing individual de-identified participant data or other relevant study documents.